CLINICAL TRIAL: NCT04089228
Title: Effects of Kinesio Taping on Upper Trapezius Trigger Points After Integrated Neuromuscular Inhibition Technique (INIT)
Brief Title: Kinesio Taping on Trapezius Trigger Points After Integrated Neuromuscular Inhibition Technique (INIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Nowal Kamran
Record Dates: First submitted 2019-09-04; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Trigger Points
Keywords: Myofascial trigger points; Kinesiotaping; Integrated Neuromuscular Inhibition Technique

STUDY DESIGN:
Who Masked: Participant
Masking Description: this study is randomized control trail, participants are randomly allocated through sealed envelope method
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape Group and INIT (Experimental): Kinesiotaping and Integrated Neuromuscular Inhibition Technique (KT + INIT )
  Interventions: Other: Kinesiotaping; Other: Integrated Neuromuscular Inhibition Technique
- INIT Group (Active Comparator): Integrated Neuromuscular Inhibition Technique (INIT)
  Interventions: Other: Integrated Neuromuscular Inhibition Technique

INTERVENTIONS:
Other: Kinesiotaping — Total of 4 sessions on upper trapezius trigger points on alternate days.
  Arms: Kinesiotape Group and INIT
Other: Integrated Neuromuscular Inhibition Technique — Sustain Pressure. Strain Counter-strain (for 90 sec) Passive Isometric Relaxation (PIR) (6-10 sec hold, 4 reps)

SUMMARY:
The aim of this research is to see the effects of kinesio taping after integrated neuromuscular inhibition technique on pain, disability, pain-pressure threshold and muscle length in patients with upper trapezius trigger points. There will be two groups experimental and control. One study group will receive kinesiotaping after integrated neuromuscular inhibition technique and the other group will only receive integrated neuromuscular inhibition technique.

DETAILED DESCRIPTION:
This study is Randomized controlled trail done at physiotherapy department of Railway General Hospital Rawalpindi. The sample size of 26 individuals calculated using open epi tool. Sampling technique applied was convenience sampling. Randomization in groups by sealed envelope method. The subjects were divided into two groups with 13 patients each. Both groups were treated with Integrated neuromuscular inhibition technique (Muscle energy Technique, sustain pressure, Strain counter-strain) while Kinesio tape was applied after INIT in only experimental group. Study duration was of 6 months. Individuals having age between 20-40 years, upper trapezius active or latent trigger points, limited side bending were included in this study. Tools used in the study were neck disability index (NDI), algometry, numeric pain rating scale (NPRS) and muscle length (side bending through inclinometer). Assessments were taken on 1st day pre and post intervention and on 4th day.

ELIGIBILITY:
Inclusion Criteria:

* Upper Trapezius Active or latent trigger points
* Limited range of motion (cervical Side Bending)

Exclusion Criteria:

* Radiculopathies
* Malignancy
* Infection
* Trauma

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 4th Day
  Changes from the baseline, The NDI is a modification of the neck disability index and it was developed by Vernon and Mior. It was designed to measure the neck pain and disability over time. It consists of 10 items, five parts sections. At the end, score is calculated by dividing the obtained score by total 50 multiplied by 100.
Pain-Pressure threshold (PPT) | 4th day
  Changes from the baseline, Pain-pressure threshold was measured with the help of an algometer.
NPRS | 4th Day
  Changes from the baseline, Numeric Pain rating scale is a scale for pain intensity starting from 0-10. Where 0 indicates no pain and 10 indicate severe pain.

SECONDARY OUTCOMES:
Muscle length measure | 4th Day
  Changes from the baseline, Muscle length of upper trapezius was measured with the help of Inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ghafoor Sajjad, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vazquez-Delgado E, Cascos-Romero J, Gay-Escoda C. Myofascial pain syndrome associated with trigger points: a literature review. (I): Epidemiology, clinical treatment and etiopathogeny. Med Oral Patol Oral Cir Bucal. 2009 Oct 1;14(10):e494-8. doi: 10.4317/medoral.14.e494. PMID 19680218
- [Background] Lluch E, Nijs J, De Kooning M, Van Dyck D, Vanderstraeten R, Struyf F, Roussel NA. Prevalence, Incidence, Localization, and Pathophysiology of Myofascial Trigger Points in Patients With Spinal Pain: A Systematic Literature Review. J Manipulative Physiol Ther. 2015 Oct;38(8):587-600. doi: 10.1016/j.jmpt.2015.08.004. Epub 2015 Sep 19. PMID 26387860
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Anesthesiol Clin. 2007 Dec;25(4):841-51, vii-iii. doi: 10.1016/j.anclin.2007.07.003. PMID 18054148
- [Background] Alvarez DJ, Rockwell PG. Trigger points: diagnosis and management. Am Fam Physician. 2002 Feb 15;65(4):653-60. PMID 11871683
- [Background] Shah JP, Gilliams EA. Uncovering the biochemical milieu of myofascial trigger points using in vivo microdialysis: an application of muscle pain concepts to myofascial pain syndrome. J Bodyw Mov Ther. 2008 Oct;12(4):371-384. doi: 10.1016/j.jbmt.2008.06.006. Epub 2008 Aug 13. PMID 19083696
- [Background] Cerezo-Tellez E, Torres-Lacomba M, Mayoral-Del Moral O, Sanchez-Sanchez B, Dommerholt J, Gutierrez-Ortega C. Prevalence of Myofascial Pain Syndrome in Chronic Non-Specific Neck Pain: A Population-Based Cross-Sectional Descriptive Study. Pain Med. 2016 Dec;17(12):2369-2377. doi: 10.1093/pm/pnw114. Epub 2016 Jun 20. PMID 28025371
- [Background] Vernon H, Schneider M. Chiropractic management of myofascial trigger points and myofascial pain syndrome: a systematic review of the literature. J Manipulative Physiol Ther. 2009 Jan;32(1):14-24. doi: 10.1016/j.jmpt.2008.06.012. PMID 19121461
- [Background] Bubnov RV. Evidence-based pain management: is the concept of integrative medicine applicable? EPMA J. 2012 Oct 22;3(1):13. doi: 10.1186/1878-5085-3-13. PMID 23088743